CLINICAL TRIAL: NCT01637415
Title: The "Prediction of Alcohol Withdrawal Severity Scale" (PAWSS): Development and Psychometric Characteristics of a New Scale for the Prediction of Complicated Alcohol Withdrawal Syndrome.
Brief Title: The "Prediction of Alcohol Withdrawal Severity Scale" (PAWSS)
Acronym: PAWSS
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jose R Maldonado, MD, Associate Professor of Psychiatry; Chief, Psychosomatic Medicine Service, Stanford University
Other Study IDs: 22731
Record Dates: First submitted 2012-06-21; First posted 2012-07-11 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Alcohol Withdrawal Syndrome
Keywords: alcohol withdrawal syndrome; prediction; severity; alcohol use disorder; complicated alcohol withdrawal; alcohol withdrawal seizures; delirium tremens; PAWSS
MeSH Terms: conditions — Alcoholism; Alcohol Withdrawal Seizures; Alcohol Withdrawal Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Although there are several tools that can be used to evaluate the severity of ongoing alcohol withdrawal syndrome (AWS), there is no available tool that can predict which patients are at risk for developing AWS at the time admission, before the patient has developed AWS. Unfortunately, there are severe symptoms of alcohol withdrawal (e.g., seizures) which may develop early in the hospitalization, and before the development of other systemic symptoms which may warn medical personnel of the possibility of impeding alcohol withdrawal (e.g., autonomic instability, delirium). The goal of this study is to evaluate the psychometric properties (e.g., predictive validity) of a new tool, the Prediction of Alcohol Withdrawal Severity Scale (PAWSS), on identifying which patients are at risk for developing complicated AWS (i.e., seizures, hallucinosis, delirium tremens) among hospitalized, medically ill patients.

DETAILED DESCRIPTION:
The investigators plan to study the psychometric properties of a new tool, the "Prediction of Alcohol Withdrawal Severity Scale" (PAWSS) on predicting the risk for the development of complicated AWS (i.e., seizures, delirium tremens) in hospitalized medically ill patients. This tool was developed through an extensive literature review which identified evidence-based predictors for AWS.

The scale consists of three portions relating to 1) an initial screening (threshold items), 2) patient's history of alcohol use and its consequences, and 3) measures of BAL and autonomic function. The investigators predict that a scale score 4 or greater will be associated with a high risk for the development of complicated AWS.

Patients will undergo examination with the PAWSS within 24 hours of hospital admission. Thereafter, all patients will undergo daily examinations with the Clinical Institute Withdrawal Assessment for Alcohol, revised (CIWA) and the Alcohol Withdrawal Severity scale (AWS scale) in order to measure the primary outcomes of the study, that is, the development and severity (i.e., moderate to severe) of AWS during the first 72-hours after admission. The study is designed to study the tool's psychometric properties including its validity and inter-rater reliability.

By providing clinicians with a tool (i.e., PAWSS) that allows them to correctly predict who will develop complicated AWS it will enable them to prophylax (i.e., preventively treat) patients at risk and thus decrease patients' morbidity and mortality, shorten length of hospital stay, minimize the significant burden on the nursing and medical staff, and improve overall patient care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients - defined as 18+ years of age
* Able to understand and communicate in English.
* Admission to the hospital within the last 24 hours to selected Stanford Hospital and Clinics inpatient units from the ED, outpatient clinics/community, or other SHC medical units.
* Without an imminent discharge plan, (within 48 hours of study screening).
* Willing and able to freely consent and participate.

Exclusion Criteria:

* Unable or unwilling to consent and participate.
* Unable to understand and communicate in English.
* Patients transferred from outside medical facilities.
* Patients with imminent discharge plan (i.e., not expected to remain in the hospital for at least 48 hours after enrollment into the study)
* Uncontrolled active seizure disorder.
* Active severe AWS (as defined by CIWA = or > 20) on initial assessment.
* Identified by the primary team as too sick to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients at Stanford Hospital and Clinics selected medical & surgical inpatient units (B2, B3, and C2), admitted directly from either Stanford ED or from any community or outpatient setting.
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Complicated alcohol withdrawal | During the first 72 hours after admission.
  Complicated withdrawal will be defined as patients meeting criteria for complicated or severe withdrawal according to DSM-IV-Tr, a CIWA-Ar score > or = to 15, or experiencing severe symptoms requiring the use of benzodiazepine agents for symptom management.

SECONDARY OUTCOMES:
Amount of benzodiazepines administered | During the first 72 hours after admission.
Transfer to ICU due to severe AWS | During the first 5 days after admission.
Development of delirium | During the first 72 hours after admission.
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Maldonado, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospitals and Clinics, Stanford, California, United States

REFERENCES:
- [Result] Maldonado JR, Sher Y, Ashouri JF, Hills-Evans K, Swendsen H, Lolak S, Miller AC. The "Prediction of Alcohol Withdrawal Severity Scale" (PAWSS): systematic literature review and pilot study of a new scale for the prediction of complicated alcohol withdrawal syndrome. Alcohol. 2014 Jun;48(4):375-90. doi: 10.1016/j.alcohol.2014.01.004. Epub 2014 Feb 19. PMID 24657098
- [Result] Maldonado JR, Nguyen LH, Schader EM, Brooks JO 3rd. Benzodiazepine loading versus symptom-triggered treatment of alcohol withdrawal: a prospective, randomized clinical trial. Gen Hosp Psychiatry. 2012 Nov-Dec;34(6):611-7. doi: 10.1016/j.genhosppsych.2012.06.016. Epub 2012 Aug 13. PMID 22898443
- [Result] Maldonado JR. An approach to the patient with substance use and abuse. Med Clin North Am. 2010 Nov;94(6):1169-205, x-i. doi: 10.1016/j.mcna.2010.08.010. PMID 20951277
- [Result] Stern TA, Gross AF, Stern TW, Nejad SH, Maldonado JR. Current approaches to the recognition and treatment of alcohol withdrawal and delirium tremens: "old wine in new bottles" or "new wine in old bottles". Prim Care Companion J Clin Psychiatry. 2010;12(3):PCC.10r00991. doi: 10.4088/PCC.10r00991ecr. No abstract available. PMID 20944765